CLINICAL TRIAL: NCT00006081
Title: A Phase II Study of Bryostatin-1 (NSC 339555) Plus Paclitaxel in Patients With Metastatic or Unresectable Locally Advanced Adenocarcinoma of the Stomach or Gastroesophageal Junction
Brief Title: Combination Chemotherapy in Treating Patients With Unresectable Locally Advanced or Metastatic Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ID99-203; U01CA070172 (NIH); P30CA016672 (NIH); MDA-ID-99203 (Other: UT MD Anderson Cancer Center); NCI-T99-0103; CDR0000068069 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2000-08-03; First posted 2003-07-25 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage III gastric cancer; stage IV gastric cancer; stage III esophageal cancer; stage IV esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Bryostatins; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bryostatin-1 + Taxol (Experimental)
  Interventions: Drug: Bryostatin-1; Drug: Paclitaxel (Taxol)

INTERVENTIONS:
Drug: Bryostatin-1 — 40 mcg/m2 one-hour infusion 24 hours after each dose of paclitaxel (i.e., day 2, 9, 16).
Drug: Paclitaxel (Taxol) — 80 mg/m^2 one-hour infusion weekly x 3 every 4 weeks
  Other Names: Taxol

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of combining bryostatin 1 and paclitaxel in treating patients who have unresectable locally advanced or metastatic stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response rate in patients with unresectable locally advanced or metastatic adenocarcinoma of the stomach or gastroesophageal junction treated with bryostatin 1 and paclitaxel.
* Determine the qualitative and quantitative toxicity and reversibility of toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 1 hour on days 1, 8, and 15 and bryostatin 1 IV over 1 hour on days 2, 9, and 16. Treatment continues every 4 weeks for at least 2 courses in the absence of disease progression or unacceptable toxicity. Patients with a complete response (CR) receive up to 4 more courses after achieving CR.

Patients are followed until death.

PROJECTED ACCRUAL: A total of 18-35 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with histologic proof of adenocarcinoma of the stomach or gastroesophageal junction will be eligible.
2. Patients must have either metastatic or unresectable local-regional cancer
3. Patients must have measurable disease, defined as lesions that can be accurately measured in at least one dimension (longest diameter to be recorded) as greater than or equal to 20 mm with conventional techniques or as greater than or equal to 10 mm with spiral CT scan.
4. Patients may not have received prior chemotherapy or immunotherapy regimen except in the adjuvant therapy that ended at least 6 months prior to registration on this study.
5. Prior limited radiation therapy is permitted. Prior radiotherapy must not have included major bone marrow containing areas (pelvis, lumbar spine), or contained the single evaluable lesion in the radiation field. A recovery period of at least 4 weeks after completion of radiotherapy is required prior to enrollment. Patients receiving chemotherapy used as radiosensitizer will not be eligible except if chemoradiotherapy was administered in the adjuvant setting (see 4.4).
6. Patients must have a life expectancy of at least 12 weeks.
7. Patients must have a performance status of less than or equal to 2 (Zubrod scale) or greater than or equal to 60% (Karnofsky scale) (see appendix B).
8. Patients must give written informed consent.
9. Acceptable liver, renal, and marrow function
10. Patients must be be at least 18 years old.
11. Patients must have recovered from recent surgery. One week must have elapsed from the time of a minor surgery and 3 weeks from major surgery.
12. This clinical trial is so designed that no person shall on the grounds of race, color, gender or national origin be excluded from participation in or be denied the benefits, or be otherwise subjected to discrimination through or under this study.

Exclusion Criteria:

1. Patients may receive no other concurrent chemotherapy, immunotherapy, or radiotherapy.
2. Patients with brain metastases are not eligible.
3. Patients with NYHA Class III or IV heart disease are not eligible (see Appendix F) as well as those patients with history of angina, myocardial infarction, or congestive heart failure within six months.
4. Pregnant or lactating women because paclitaxel and bryostatin-1, like most other anticancer agents, may be harmful to the developing fetus and nursing newborn or infant. All women of child-bearing potential must have a negative pregnancy test prior to entry into the study. All patients of child-bearing potential must be advised of the importance of avoiding pregnancy and using appropriate methods of contraception while participating in this investigational trial.
5. Patients with serious intercurrent infections, or nonmalignant medical illnesses that are uncontrolled or whose control may be jeopardized by the complications of this therapy, are ineligible.
6. Patients with psychiatric disorders rendering them incapable of complying wiht the requirements of the protocol are ineligible.
7. Patients with serum calcium greater > 12 mg/dl or symptomatic hypercalcemia under treatment are ineligible.
8. Patients with only bone metastases.
9. Patients with any concurrent active malignancy other than non-melanoma skin cancers or carcinoma-in-situ of the cervix. Patients with previous malignancies but without evidence for greater than or equal to 5 years will be allowed to enter the trial.
10. Patients wit bleeding diathesis or those requiring anticoagulation will be excluded.
11. Patients with only non-measurable disease, defined as all other lesions, including small lesions (longest diameter < 20 mm with conventional techniques or < 10 mm with spiral CT scan) and truly non-measurable lesions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2000-06; Primary Completion 2005-09 (Actual); Study Completion 2005-09 (Actual)

PRIMARY OUTCOMES:
Number of Patients with Response after 2 Cycles of Treatment | 8 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jaffer A. Ajani, MD, Study Chair — M.D. Anderson Cancer Center
Locations (2):
- United States (2):
  - CCOP - M.D. Anderson Research Base, Houston, Texas
  - University of Texas - MD Anderson Cancer Center, Houston, Texas

REFERENCES:
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org